CLINICAL TRIAL: NCT03414788
Title: PHASE 1B, OPEN LABEL STUDY TO CHARACTERIZE THE DISTRIBUTION OF A SINGLE INTRAVENOUS DOSE OF [124I]-IODOBENZOYL (IB)-PF-06687234 WITH CONCURRENT ADMINISTRATION OF NON-RADIOLABELED PF-06687234 AS ASSESSED WITH POSITRON EMISSION TOMOGRAPHY AND COMPUTED TOMOGRAPHY (PET-CT) IMAGING IN MODERATE TO SEVERE ULCERATIVE AND CROHN'S COLITIS SUBJECTS
Brief Title: Distribution of a Single IV Dose Of [124I]-Pf 06687234 and Pf 06687234 Assessed With PET-CT Imaging In Moderate To Severe Ulcerative Colitis and Crohn's Disease
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn due to not being able to recruit subjects.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B7581003
Record Dates: First submitted 2018-01-08; First posted 2018-01-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Inflammatory Bowel Disease
Keywords: Positron Emission Tomography (PET), Inflammatory Bowel Disease, Safety, PKPlasma
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm - PF 06687234 and [124I]IB PF 06687234 (Experimental): PF 06687234 and [124I]IB PF 06687234
  Interventions: Biological: PF 06687234; Biological: [124I]IB PF 06687234

INTERVENTIONS:
Biological: PF 06687234 — Subjects will be given single, intravenous dose of PF 06687234 and [124I]IB PF 06687234 simultaneously
Biological: [124I]IB PF 06687234 — Subjects will be given single, intravenous dose of PF 06687234 and [124I]IB PF 06687234 simultaneously

SUMMARY:
The purpose of the study is to evaluate the PK, safety and tolerability of PF-06687234 and [124I]IB-PF-06687234 (simultaneously given) in subjects with moderate to severe Ulcerative Colitis or Crohn's Disease. The study used PET-CT scan imaging to assess the distribution of PF-06687234 and [124I]IB-PF-06687234 over 24 and 72 hours in colon (inflamed and non-inflamed), plasma, colon, liver, spleen, kidney and small intestine.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female subjects of non-child bearing potential, 18 years to 75 years of age inclusive at the time of informed consent
* Only women of non-child bearing potential
* Diagnosis of active UC (histologic) or CD prior to study entry for a minimum of 4 months
* Subjects with moderate to severe, active UC as defined by Mayo endoscopic index of at least 2; or subjects with moderate to severe, active CD as defined by SES-CD score of at least 7.

Exclusion Criteria:

* Clinically significant/unstable clinical conditions (eg. cancer hematological, endocrine etc)
* Active enteric infections
* Other forms of colitis such as infectious colitis etc

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-07 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Percent injected radioactivity dose per kilogram (% ID/kg) in the colon (inflamed and non inflamed) and plasma | 24 hours
  Treatment Arm
Standardized uptake value (SUV) in the colon (inflamed and non inflamed) | 24 hours
  Treatment Arm

SECONDARY OUTCOMES:
AUC of PF 06687234 plasma concentrations over time | 42 days
  Treatment Arm
AUC of plasma radioactivity concentration (% ID/kg) | 24 hours
  Treatment Arm
AUC in plasma, colon, liver, spleen, kidney and small intestine | 24 hours
  Treatment Arm
Ratio of radioactivity AUC0-24H between colon, liver, spleen, kidney and small intestine to plasma | 24 hours
  Treatment Arm
Frequency of clinically relevant abnormalities for Safety Labs | 42 days
  Treatment Arm
Cmax of PF 06687234 plasma concentrations over time | 42 days
  Treatment Arm
Tmax of PF 06687234 plasma concentrations over time | 42 days
  Treatment Arm
Cmax of plasma radioactivity concentration (% ID/kg) | 24 hours
  Treatment Arm
Tmax of plasma radioactivity concentration (% ID/kg) | 24 hours
  Treatment Arm
Cmax of radioactivity in plasma, colon, liver, spleen, kidney and small intestine | 24 hours
  Treatment Arm
Tmax of radioactivity in plasma, colon, liver, spleen, kidney and small intestine | 24 hours
  Treatment Arm
Frequency of clinically relevant abnormalities for vital signs | 42 days
  Treatment Arm
Frequency of clinically relevant abnormalities for ECG | 42 days
  Treatment Arm
Frequency of clinically relevant abnormalities for Immunogenicity | 42 days
  Treatment Arm

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7581003